CLINICAL TRIAL: NCT03963778
Title: A Study Investigating the Impact of Organisational Culture on Nutritional Care in Hospitalised Patients
Brief Title: Organisational Culture and Nutritional Care
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1718/IRASGY/1
Record Dates: First submitted 2019-05-10; First posted 2019-05-28 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Nutrition
Keywords: Malnourishment; Nutritional Deficiency; Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Improving nutritional care — The interventions will be co-designed with the action research team

SUMMARY:
The study explores the impact of organisational culture on multidisciplinary teams in the provision of nutritional care for older hospitalised acute in-patients by collaborating with patients and/or their relatives and healthcare practitioners to influence change.

DETAILED DESCRIPTION:
This study adopts an action research (AR) approach given that sustained change is more likely if it incorporates authentic staff engagement. The key choice made in formulating the research design is to adopt an approach that is collaborative and participatory in a process of action and learning.

Here, eligible health practitioners involved in any aspect of the patients' food and nutritional care or helping to feed patients during mealtimes would be represented in one central team, engaging as co-researchers in the study.

Patients and/or relatives will participate in a focus group or interview session. The AR team participants will be involved in the iterative action research cycle, reflecting on current nutritional care practices, collectively evaluate patients' stories and consider ways to improve eating and drinking on the wards. The AR team will meet throughout the course of 12 months.

The study will provide insight into the impact of organisational culture ('the way the investigators do things') in the delivery of good nutritional care and elucidate the roles and responsibilities of nurses and other staff groups involved in the provision of nutritional care.

This research will provide data on the organisational culture of interdisciplinary teams working at both micro and macro levels while providing insight into the potential for AR to be used in a wider arena within the hospital to improve practice.

ELIGIBILITY:
Inclusion Criteria:

* Recently discharged patients aged 65 or over
* Recently discharged patients at the time of data collection
* Who at the time of admission received oral nutrition and hydration

Exclusion Criteria:

* Patients aged under 65
* Current in-patients
* Patients who have had no oral nutrition. e.g patients who had Percutaneous Endoscopic Gastrostomy (PEG) feeds whilst admitted
* Patients who are feeling too unwell to participate
* Patients lacking the mental capacity to give verbal or written consent

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Recently discharged patients from an acute healthcare setting.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Focus Group sessions / Action research team meetings | 12 months
  The action research team will have focus group/meetings involving health professionals willing to participate as co-researchers to collectively draw on their experiences to collaborate and implement interventions to improve nutritional care delivery for patients following the iterative AR cycles; planning, taking action, observing and evaluating interventions. The group meetings will be spread across 12 months.
  Outcome measures are obtained from interventions implemented as agreed by the team and as informed by preliminary data (such as the Malnutrition Universal Screening Tool ('MUST') audit).

SECONDARY OUTCOMES:
Interview/focus group | 8 months
  Semi-structured interview or focus group with patients and /or their relatives willing to share their experiences on food and nutritional care.
Malnutrition Universal Screening Tool Hospital Audit. | 18 months
  Evaluation of 'MUST' Audit pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Scammell, PhD, Study Director — Associate Professor
Locations (1):
- Bournemouth University, Bournemouth, Dorset, United Kingdom